CLINICAL TRIAL: NCT03116061
Title: The Frequency of Family Physician Visits and the Extent of Family Difficulties Reported by Family Physicians Appear to be Decompensation Risk Factors for Multimorbid Outpatients in a Primary Care Feasibility Study
Brief Title: The Reported Frequency of FP Visits and Family Difficulties Should Alert FPs and Help Them to Prevent Severe Outcomes in Multimorbid Outpatients
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: ERCR SPURBO (Other)
Responsible Party: Sponsor
Other Study IDs: SPURBO
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Multimorbidity
Keywords: Multimorbidity; Family Medicine; decompensation; predictive value
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multimorbidity cohort: The study population included a random sample of multimorbid patients (according to the EGPRN definition of multimorbidity). Patients were selected by 19 FPs in their offices in the county of Finistere (in north-west France) from July 2014 to December 2014. Randomization was achieved by including the first four multimorbid patients (according to the inclusion criteria) encountered during their second working day of each week. As patients were booking their appointments with the practice without the FPs' clearance, the FPs were not able to select them
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — This questionnaire was to explore potential decompensation risk factors within themes and subthemes of multimorbidity

SUMMARY:
The European General Practitioners Research Network (EGPRN) designed and validated a comprehensive definition of multimorbidity using a systematic literature review and qualitative research throughout Europe. This definition was tested as a model to assess decompensation in multimorbid outpatients.

The objective is to assess which criteria in the EGPRN concept of multimorbidity could detect decompensating outpatients in a primary care cohort at a 6-month follow-up and to assess whether a large scale cohort with FPs would be feasible.

DETAILED DESCRIPTION:
Method: Family Physicians included a random sample of multimorbid patients who attended appointments in their offices from July to December 2014. Inclusion criteria were those of the EGPRN definition of Multimorbidity. Exclusion criteria were patients under legal protection and those unable to complete the 2-year follow-up. Decompensation was defined as the occurrence of death or hospitalization for more than seven days. Statistical analysis was undertaken with uni- and multivariate analysis at a 6-month follow-up using a combination of approaches including both automatic classification and expert decision making. A Multiple Correspondence Analysis (MCA) confirmed results consistency and completed the process with a projection of illustrative variables. A logistic regression was finally performed in order to identify and quantify risk factors for decompensation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were patients meeting the criteria for the definition of multimorbidity according to the EGPRN definition: any combination of chronic disease with at least one other disease (acute or chronic) or a bio psychosocial factor (associated or not) or a somatic risk factor.

Exclusion Criteria:

* Exclusion criteria were patients not meeting the criteria of the definition of multimorbidity, the inability to follow the study over time (known to be leaving the practice in the following months), patients under legal protection, outpatients in palliative care for whom survival was estimated by the FPs at less than three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included a random sample of multimorbid patients (according to the EGPRN definition of multimorbidity). Patients were selected by 19 FPs in their offices in the county of Finistere (in north-west France) from July 2014 to December 2014.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To detect the decompensating outpatients | 6 months
  To assess which criteria in the EGPRN concept of multimorbidity could detect decompensating outpatients in a primary care cohort at a 6-month follow-up and to assess whether a large scale cohort with FPs would be feasible

IPD SHARING:
Plan to Share IPD: No